CLINICAL TRIAL: NCT05718817
Title: A Multicenter, Open-label, Long-term, Safety, Tolerability, and Efficacy Study of XEN1101 in Subjects Diagnosed With Epilepsy
Brief Title: An Open-label Study of XEN1101 in Epilepsy
Acronym: X-TOLE4
Status: Enrolling by invitation | Phase: Phase 3 | Type: Interventional
Sponsor: Xenon Pharmaceuticals Inc. (Industry)
Collaborators: Worldwide Clinical Trials (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XPF-010-304; 2022-502282-24-00 (EU CTIS Number)
Record Dates: First submitted 2023-01-13; First posted 2023-02-08 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Focal Epilepsy; Tonic-Clonic Seizures
Keywords: Epilepsy; Seizures
MeSH Terms: conditions — Epilepsies, Partial; Seizures; Epilepsy | interventions — XEN1101

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- XEN1101 15 or 25 mg/day (Experimental): XEN1101 15 or 25 mg/day
  Interventions: Drug: XEN1101

INTERVENTIONS:
Drug: XEN1101 — XEN1101 capsules
  Other Names: Azetukalner

SUMMARY:
This study will evaluate the long term safety, tolerability, pharmacokinetics (PK), and efficacy of XEN1101 in subjects with Focal Onset Seizures (FOS) or Primary Generalized Tonic-Clonic Seizures (PGTCS) for the treatment of seizures for up to 3 years.

DETAILED DESCRIPTION:
This is an Open Label Extension study of the following Phase 3 clinical studies: XPF-010-301 (X-TOLE2), XPF-010-302 (X-TOLE3), and XPF-010-303 (X-ACKT). This study will evaluate the long-term safety, tolerability, PK, and efficacy of XEN1101 in subjects with FOS or PGTCS for the treatment of seizures for up to 3 years. Subjects who successfully completed and did not terminate early from one of the antecedent studies (X-TOLE2, X-TOLE3, or X-ACKT) are eligible to participate in X-TOLE4.

Following enrollment into X-TOLE4, subjects will undergo a treatment period of up to 3 years, during which there will be a visit at 2-, 4-, and 13-weeks post-entry, with subsequent visits occurring at 13-week intervals during the first year, and then at 26-week intervals (with a telephone call in between) until dosing is completed.

Subjects will be initially assigned to XEN1101 as follows:

* 25 mg QD for subjects aged ≥18 years
* For subjects aged ≥12 and <18 years

  * 15 mg QD for those

    * who weigh <45 kg at the start of the X-TOLE4 study
    * who weighed <45 kg during the X-ACKT study
    * who weighed ≥45 kg at randomization in the X-ACKT study and had dose reduction(s) for intolerability
  * 25 mg QD for all others

Subjects will be instructed to orally take XEN1101 once daily (QD) with an evening meal. Subjects will be expected to keep a daily seizure eDiary with a minimum of 80% compliance for the duration of the extension study (reporting on ≥80% of days between visits).

Upon completion of dosing at the end of the treatment period, there will be an 8-week follow up period.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be properly informed of the nature and risks of the study and give informed consent in writing prior to entering the study (for adult subjects) and for adolescent subject's parent/legal guardian and subject gives informed consent or assent in writing prior to entering the study.
2. Subject must have successfully completed the double-blind treatment period (DBP) and have not terminated early from Study X-TOLE2, X-TOLE3, or X-ACKT, met all eligibility requirements, and had no important protocol deviations (in the opinion of the sponsor) or adverse events (AEs) (in the opinion of the investigator) that would preclude the subject's entry into the long-term extension study.
3. In the opinion of the investigator, the subject is able to understand verbal and written instructions and will adhere to all study schedules and requirements.
4. Subject is able to keep accurate seizure diaries.

Exclusion Criteria:

1. Subject met any of the withdrawal criteria while in Study X-TOLE2, X-TOLE3, or X-ACKT.
2. Subject has any medical condition, personal circumstance, or ongoing AE (from Study X-TOLE2, X-TOLE3, or X-ACKT) that, in the opinion of the investigator, exposes the subject to unacceptable risk by participating in the study, or prevents adherence to the protocol.
3. Subject is planning to enter a clinical study with a different investigational drug or planning to use any experimental device for treatment of epilepsy or any other medical condition during the study and until 28 days after completion of this study.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 880 (Estimated)
Dates: Start 2023-04-25 (Actual); Primary Completion 2028-07 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
The adverse events | From the start of treatment in the open-label extension (OLE) study through 8 weeks after the last dose.
  To assess the safety and tolerability of XEN1101

SECONDARY OUTCOMES:
Change in monthly seizure rate | From baseline through the active extension treatment (Week 156).
  Percent change in monthly seizure rate recorded at baseline (in the antecedent studies) compared to each 4-week assessment period in the treatment period in X-TOLE4.
Proportion of responders | From baseline through the active extension treatment (Week 156).
  Proportion of responders (subjects experiencing ≥50% reduction in seizure frequency from baseline) in each consecutive 4-week assessment period of the treatment period of the OLE study.
Change in Clinical Global Impression of Severity (CGI-S) | From baseline through the active extension treatment (Week 156).
  Improvement in Clinical Global Impression of Severity (CGI-S) scores over time.
Change in Patient Global Impression of Severity (PGI-S) | From baseline through the active extension treatment (Week 156).
  Improvement in Patient Global Impression of Severity (PGI-S) scores over time.
Change in Quality of Life in Epilepsy Inventory (QOLIE-31) | From baseline through the active extension treatment (Week 156).
  Change in the 31-Item Quality of Life in Epilepsy Inventory (QOLIE-31) over time.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Xenon Pharmaceuticals Inc.
Locations (145):
- United States (52):
  - Xenoscience, Phoenix, Arizona
  - University of Arizona - Health Sciences, Tucson, Arizona
  - Clinical Trials, Inc, Little Rock, Arkansas
  - Brain Science Research Institute, Los Angeles, California
  - UC Irvine Health, Orange, California
  - University of California, Davis Clinical & Translational Science Center Clinical Research (CCRC), Sacramento, California
  - University of Colorado Hospital Anschutz Outpatient Pavilion, Aurora, Colorado
  - Mayo Clinic Florida, Jacksonville, Florida
  - Serenity Research Center, LLC, Miami, Florida
  - Research Institute of Orlando, LLC, Orlando, Florida
  - Panhandle Research & Medical Clinic, Pensacola, Florida
  - University of South Florida, Tampa, Florida
  - Encore Medical Research of Weston, LLC, Weston, Florida
  - Hawaii Pacific Neuroscience, Honolulu, Hawaii
  - Consultants in Epilepsy and Neurology, Boise, Idaho
  - Indiana University School of Medicine, Indianapolis, Indiana
  - The University of Kansas Medical Center, Kansas City, Kansas
  - Bluegrass Epilepsy Research, LLC, Lexington, Kentucky
  - Kentucky Clinic, Lexington, Kentucky
  - MMP Neurology, Scarborough, Maine
  - University of Maryland Medical Center, Baltimore, Maryland
  - Mid-Atlantic Epilepsy and Sleep Center, Bethesda, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - UMass Chan Medical School, Worcester, Massachusetts
  - University of Michigan Hospitals, Ann Arbor, Michigan
  - Wayne State University, Detroit, Michigan
  - Michigan State University, East Lansing, Michigan
  - Cornwell Health (Spectrum Health Hospitals), Grand Rapids, Michigan
  - Minneapolis Clinic of Neurology, Burnsville, Minnesota
  - Saint Louis University Medical School, St Louis, Missouri
  - Northeast Epilepsy Group, Hackensack, New Jersey
  - Dent Neurosciences Research Center, Buffalo, New York
  - New York University Comprehensive Epilepsy Center, New York, New York
  - Mount Sinai Health, New York, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - Montefiiore Medical Center, The Bronx, New York
  - Onsite Clinical Solutions, Charlotte, North Carolina
  - Duke University, Durham, North Carolina
  - Meridian Clinical Research, LLC, Raleigh, North Carolina
  - Summa Health, Akron, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Providence Neurological Specialities, Portland, Oregon
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Austin Epilepsy Care Center, Austin, Texas
  - ANESC Research, El Paso, Texas
  - UT Health San Antonio, San Antonio, Texas
  - University of Utah Clinical Neurosciences Center, Salt Lake City, Utah
  - Carilion Clinic, Roanoke, Virginia
  - Sentara Neurology Specialists, Virginia Beach, Virginia
  - University of Washington Main Hospital, Seattle, Washington
  - Aurora St. Luke's Medical Center, Milwaukee, Wisconsin
- Argentina (10):
  - Hospital General de Agudos "José M. Ramos Mejía", Buenos Aires
  - Asociacion Medica de Lomas de Zamora S.A. - Policlinicio Lomas, Buenos Aires
  - STAT Research S.A., Buenos Aires
  - Centro de Psicología Médica San Martín de Tours SRL (CITES-INECO), Buenos Aires
  - Hospital Italiano de Buenos Aires, Buenos Aires
  - CENyR, Centro de Especialidades Neurologicas u Rehabilitacion, Buenos Aires
  - FLENI (Fundación para la Lucha contra las Enfermedades Neurológicas de la Infancia), Buenos Aires
  - Hospital Córdoba, Córdoba
  - Hospital De Alta Complejidad en Red El Cruce - Dr Nester Carlos Kirchner Servicio de Atencion Medica Integral Para la Communidad, San Juan Bautista
  - Sanatorio del SUR S.A., San Miguel de Tucumán
- Australia (9):
  - Prince of Wales Hospital, Randwick, New South Wales
  - Royal Prince Alfred Hospital, Camperdown
  - St Vincent's Hospital Melbourne, Fitzroy
  - Austin Health Pharmacy Clinical Trials, Heidelberg
  - Southern Neurology, Kogarah
  - Alfred Hospital Neurology CT Dept of Neuroscience, Melbourne
  - The Royal Melbourne Hospital, Parkville
  - Mater Misericordiae Ltd South Brisbane, South Brisbane
  - Westmead Hospital Dept. of Neurology Epilepsy Unit, Westmead
- Austria (2):
  - University Hospital Innsbruck, Innsbruck
  - Universitatsklinik fur Neurologie, Medizinische Universitat Wien, Vienna
- Belgium (2):
  - Cliniques Universitaires Saint-Luc (UCL), Brussels
  - Universitair Ziekenhuis Gent, Ghent
- Bulgaria (2):
  - Hospital for active treatmnt Puls AD Neurology Dpt, Blagoevgrad
  - MHATNP St. Naum, Sofia
- Canada (3):
  - Center for Neurologic Research, Lethbridge, Alberta
  - London Health Sciences Center, London, Ontario
  - Le Centre Hospitalier de l'Universite' de Montreal (CHUM), Montreal
- Chile (2):
  - Centro de investigación Clinica UC, Santiago
  - Hospital Clinico Viña del Mar, Viña del Mar
- Croatia (3):
  - Altavita Centar j.d.o.o., Zagreb
  - Poliklinika Bonifarm, Zagreb
  - University Hospital Centre Zagreb, Zagreb
- Czechia (2):
  - Motol University Hospital, Prague
  - Forbeli s.r.o., Prague
- France (5):
  - Hopital Neurologique Pierre Wertheimer, Hospices Civils de Lyon, Lyon
  - Hôpital Fondation Adolphe de Rothschild, Paris
  - Hôpitaux Universitaires Pitié Salpêtrière, Paris
  - CHU De Rennes - Hôpital Pontchaillou, Rennes
  - Hôpital de Hautepierre, Strasbourg
- Georgia (2):
  - American Hospital Network LLC, Tbilisi
  - Institute of Neurology and Neuropsychology, Tbilisi
- Germany (7):
  - Universitätsklinikum Aachen, Aachen
  - Krankenhaus Mara gGmbH, Bielefeld
  - Universitätsklinikum, ZNN - Epilepsiezentrum Frankfurt Rhein-Main, Frankfurt
  - University Hospital Freiburg, Freiburg im Breisgau
  - Philipps-Universität Marburg, Marburg
  - Klinikum der Universität München, München
  - Universitaets-Und Rehabilitations Ulm (RKU), Ulm
- Semmelweis Egyetem, Idegsebeszeti es Neurointervencios Klinika, Budapest, Hungary
- Beaumont Hospital, Dublin, Ireland
- Israel (3):
  - Hadassah Medical Center (HMC), Jerusalem
  - Kaplan Medical Center (KMC), Rehovot
  - The Tel Aviv Sourasky Medical Center, Tel Aviv
- Italy (4):
  - IRCCS Istituto delle Scienze Neurologiche Bologna, Bologna
  - Universita' Degli Studi Gabriele d'Annunzio Di Chieti, Chieti
  - Azienda Ospedaliero Universitaria Pisana, Pisa
  - Azienda Ospedaliero Universitaria Policlinico Umberto I, Roma
- Mexico (3):
  - Human Science Research Trials, Mexico City
  - Grupo Medico Camino SC, Mexico City
  - Neurociencias Estudios Clínicos SC, Sinaloa
- New Zealand (2):
  - University of Auckland, Auckland
  - Waikato Hospital, Hamilton
- Poland (6):
  - Centrum Medyczne Neuromed, Bydgoszcz
  - COPERNICUS Podmiot Leczniczy Sp. z o.o., Gdansk
  - NZOZ Neuromed M. i M., Lublin
  - Twoja Przychodnia Nowosolskie Centrum Medyczne, Nowa Sól
  - MTZ Clinical Research Powered by Pratia, Warsaw
  - Neurosphera Sp z o.o., Warsaw
- Portugal (7):
  - Centro Hospitalar Universitário de Coimbra (CHUC), Coimbra
  - Hospital Senhora da Oliviera de Guimaraes, Guimarães
  - Centro Hospitalar Lisboa Ocidental, EPE - Hospital Egas Moniz, Lisbon
  - Centro Hospitalar Universitario de Santo António, E.P.E, Porto
  - Unidade Local de Saúde de São João, Porto
  - Unidade Local Saúde Matosinhos, Porto
  - Centro Hospitalar de Entre o Douro e Vouga, Santa Maria da Feira
- Spain (10):
  - Hospital Universitario Cruces, Barakaldo
  - Vall d'Hebron Hospital, Barcelona
  - Hospital Vithas La Milagrosa, Madrid
  - Hospital Ramón Y Cajal, Madrid
  - Hospital Ruber Internacional, Madrid
  - Hospital Clinico San Carlos, Madrid
  - Hospital Universitario Fundación Jiménez Díaz, Madrid
  - Hospital Regional De Malaga, Málaga
  - Hospital La Fe, Valencia
  - Hospital Clinico Universitario de Valladolid, Valladolid
- United Kingdom (7):
  - Leeds Teaching Hospitals NHS Trust, Leeds, England
  - Cardiff and Vale UHB, Cardiff, Wales
  - Queen Elizabeth Hospital Birmingham, Birmingham
  - St George's Hospital NHS Foundation Trust, London
  - University College London, London
  - John Radcliffe Hospital, Oxford
  - Salford Royal NHS Foundation Trust - Greater Manchester Neuroscience Centre (GMNC), Salford

IPD SHARING:
Plan to Share IPD: No